CLINICAL TRIAL: NCT03123861
Title: Randomized Controlled Trial of Gabapentin Versus Placebo for Postoperative Pain After Sacrospinous Ligament Fixation for Pelvic Organ Prolapse
Brief Title: Gabapentin for Postop Pain After SSLF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16-3392
Record Dates: First submitted 2017-03-26; First posted 2017-04-21 (Actual); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-09

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; postoperative gluteal pain; opioid use
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Active Comparator): Participants will take 300 mg Gabapentin for the first 3 days after surgery, then dose escalate to 300 mg twice a day (BID) for an additional 11 days.
  Interventions: Drug: Gabapentin
- Placebo oral capsule (Placebo Comparator): Participants will take placebo for the 2 weeks after surgery.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Gabapentin — Patients randomized to this arm will receive 2 weeks of gabapentin post-operatively.
  Other Names: neurontin
  Arms: Gabapentin
Drug: Placebo oral capsule — Patients randomized to this arm will receive 2 weeks of placebo post-operatively..
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
Purpose: To assess the impact of gabapentin versus placebo on overall postoperative pain and gluteal pain at 7 days after vaginal sacrospinous ligament suspension for apical pelvic organ prolapse.

Participants: English-speaking women planning to undergo a vaginal SSLF. Concurrent procedures can be performed except total vaginal hysterectomy, colpocleisis, anal sphincteroplasty, fistula surgery, or urethral diverticulectomy

Procedures (methods): Patients will be randomized to receive either 2 weeks of gabapentin or placebo for 2 weeks post-operatively. Standard of care pain medications will be given to both groups. Patients will be followed for 6 weeks post-operatively.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP), the herniation of the bladder, uterus, or rectum, into and often beyond, the vaginal opening, affects 40% of postmenopausal women and significantly impairs quality of life. POP is often managed surgically, and currently, one in every eight women will undergo POP surgery during her lifetime.

A commonly performed procedure for POP is a sacrospinous ligament fixation (SSLF), which is a vaginal surgery that involves suspending the vaginal apex to the sacrospinous ligament suspension with sutures. Beyond routine postoperative pain, a sacrospinous ligament fixation may result in significant gluteal pain as a result of the vaginal sutures affecting/impinging on the sacral nerve roots. Unfortunately, postoperative gluteal pain is not uncommon with 12% of patients reporting significant gluteal pain and 4% having persistent pain 6 weeks after surgery.

This study aims to compare the impact of gabapentin versus placebo on postoperative pain after SSLF. The rationale is that studies have shown that preoperative gabapentin, a non-opioid analgesic, resulted in a lower narcotic use postoperatively. Decreasing the use of standard of care postoperative narcotic pain medications would also decrease adverse events due to narcotics such as nausea, vomiting, and constipation, and potentially decrease the long-term risk of opioid dependence. As an additional benefit, a careful assessment of actual opioid will help to inform best practices for prescribing, as we may be overprescribing narcotic medications for this type of surgery. This study will evaluate a longer two-week course of gabapentin because it is currently standard of care to use gabapentin to treat neuropathic pain after SSLF; thus, gabapentin may help to address overall pain as well as neuropathic gluteal pain that can occur after SSLF. Furthermore, gabapentin is a relatively safe medication with the primary adverse events being dizziness and sedation.

Given the risk of overall postoperative pain and neuropathic gluteal pain after a sacrospinous ligament fixation for POP and the evidence that perioperative gabapentin may decrease acute pain and neuropathic pain, this study proposes a novel randomized trial to compare perioperative gabapentin versus placebo on postoperative pain after a vaginal SSLF surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18+
* English-speaking
* Planning to undergo a vaginal SSLF

Exclusion Criteria:

* Pregnant or planning to become pregnant during study participation
* Prior vaginal mesh surgery for pelvic organ prolapse
* Planning a concurrent total vaginal hysterectomy, colpocleisis (total vaginectomy or LeFort colpocleisis), mesh excision, anal sphincteroplasty, fistula repair, or urethral diverticulectomy
* Cognitive impairment (indicated by a score of 0-2 on Mini-Cog)
* Currently taking gabapentin or pregabalin (Lyrica) or previous intolerance to gabapentin or pregabalin
* Daily use of narcotics for ≥ 2 months
* Acute or chronic renal failure based on past medical history (PMH) or glomerular filtration rate (GFR) < 30ml/min (see meds info below)
* Severe uncontrolled depression or bipolar disease based on PMH
* Fall risk if history of fall in last year or current use of cane/walker

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wu, MD, MPH, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu JM, Dieter AA, Feliciano KM, Geller EJ, Willis-Gray M. Randomized Clinical Trial of Gabapentin Versus Placebo for Pain After Sacrospinous Ligament Fixation. Female Pelvic Med Reconstr Surg. 2022 Feb 1;28(2):65-71. doi: 10.1097/SPV.0000000000001064. PMID 35084369

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gabapentin | Placebo Oral Capsule
Started | 22 | 23
Received Intervention | 21 | 22
Completed | 19 | 20
Not Completed | 3 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Gabapentin: Participants will take 300 mg Gabapentin for the first 3 days after surgery, then dose escalate to 300 mg BID for an additional 11 days.
  Gabapentin: Patients randomized to this arm will receive 2 weeks of gabapentin post-operatively.
- Total: Total of all reporting groups
Arm/Group | Gabapentin | Placebo Oral Capsule | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (7.8) | 61.2 (13.7) | 62.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 0 | 2 | 2
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 23 | 45
Body Mass Index [Mean (Standard Deviation); unit: kg / m^2] | 29.1 (4.6) | 28.1 (4.1) | 28.6 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Pain During Normal Activities (Surgical Pain Scale Item 2)
Description: Post-operative pain at week 1 will be measured by item 2 of the surgical pain scale (SPS). This item asks for the average amount of pain felt during normal activity in the last 24 hours on a scale of 1-10 with 10 representing the most intense/worst pain.
Time Frame: 7 days after surgery
Population: Participants who underwent sacrospinous ligament fixation surgery with follow-up data 7 days after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 19 | 20
units on a scale | 1.6 (1.5) | 3.2 (2.6)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo Oral Capsule; Test type: Superiority; p = 0.09, t-test, 2 sided

2. Secondary Outcome: Gluteal Pain During Normal Activities
Description: Gluteal post-op pain will be measured by an item similar to that used for the primary outcome which asks for the average amount of gluteal pain felt during normal activity in the last 24 hours on a scale of 1-10 with 10 representing the most intense/worst pain.
Time Frame: 7 days after surgery
Population: Participants who underwent a sacrospinous ligament fixation surgery with follow-up data 7 days after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 19 | 20
units on a scale | 2.1 (2.0) | 3.4 (2.4)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo Oral Capsule; Test type: Superiority; p = 0.09, t-test, 2 sided

3. Secondary Outcome: Worst Pain (Surgical Pain Scale Item 4)
Description: Post-operative pain will be measured by item 4 of the surgical pain scale (SPS). This item asks for how unpleasant or disturbing the worst pain was in the last 24 hours on a scale of 1-10 with 10 representing the most intense/worst pain
Time Frame: 7 days after surgery
Population: Participants who underwent sacrospinous ligament fixation surgery with follow-up data 7 days after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 19 | 20
units on a scale | 2.4 (2.4) | 4.0 (2.7)
Statistical Analysis 1: Comparison: Gabapentin vs Placebo Oral Capsule; Test type: Superiority; p = 0.08, t-test, 2 sided

4. Secondary Outcome: Daily Narcotic Use
Description: Median daily post-op narcotic pain medication in morphine milliequivalents per day during the first 14 days after surgery
Time Frame: First 14 days after surgery
Population: Participants who underwent sacrospinous ligament fixation surgery with follow-up data 7 days after surgery
Measure: Median (Inter-Quartile Range); unit: morphine milliequivalents per day
Arm/Group | Gabapentin | Placebo Oral Capsule
Number analyzed (Participants) | 19 | 20
morphine milliequivalents per day | 1.6 [0.5 to 4.4] | 1.6 [0.4 to 5.5]
Statistical Analysis 1: Comparison: Gabapentin vs Placebo Oral Capsule; Test type: Superiority; p = 0.91, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From the day of surgery until the 6-week postoperative visit
Arm/Group | Gabapentin | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 2/21 | 0/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gabapentin (N=21) | Placebo Oral Capsule (N=22)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT03123861/Prot_SAP_000.pdf